CLINICAL TRIAL: NCT01738971
Title: Pharmacy Based Interventions for Initiating Effective Contraception Following the Use of Emergency Contraception : a Feasibility Study
Brief Title: Initiating Contraception After Emergency Contraception From Pharmacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Protocol ECfe03; 182. (Other: Edinburgh and Lothians Health Foundation)
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Results first posted 2014-08-18 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Contraceptive Use After Emergency Contraception
Keywords: emergency contraception; community pharmacy
MeSH Terms: interventions — Levonorgestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- control (standard care) (No Intervention): standard verbal and written advice on contraception from pharmacy
- rapid access (Experimental): rapid access to family planning service
  Interventions: Other: rapid access
- progestogen only pill (Experimental): one month progestogen only pill
  Interventions: Other: one month progestogen only pill

INTERVENTIONS:
Other: rapid access — Provision of box which the participant can take to local family planning clinic (contraceptive service) allowing rapid access (i.e. will be seen by a health professional for a consultation regarding contraception there and then).
  Arms: rapid access
Other: one month progestogen only pill — Provision of 1 month supply of a progestogen only pill (levonorgestrel 35mcg - Norgeston, Bayer, UK)
  Other Names: Norgeston (Bayer, UK)
  Arms: progestogen only pill

SUMMARY:
Pharmacists do not provide immediate contraception to women after emergency contraception (EC); they can only give advice on local contraceptive services.

The investigators wish to establish the following 2 pharmacy- based interventions in NHS Lothian, designed to increase uptake of effective contraception as soon as possible, after EC

1. Pharmacists would provide one packet of progestogen-only pills, giving women one month to arrange an appointment with contraceptive services.
2. Rapid access to a family planning clinic upon presentation of the empty EC packet. Women would be seen as a 'walk-in' and contraception provided.

If feasible, these interventions could reduce unintended pregnancies.

Participating pharmacies will be randomised to provide one of the interventions, or standard care (verbal/written advice on local contraceptive services).

Women requesting EC from study pharmacies will be recruited by the research nurse/doctor to participate in the study that will involve them consenting to contact by telephone 6-8 weeks after EC by the researcher, to evaluate the interventions in terms of :

(i) determine women's experiences/ views of the interventions and control. (ii) determine if women have commenced effective contraception and if not , reasons why.

A subset of 12 women will also be invited for in-depth interview to collect more detailed qualitative data on their EC experience.

The investigators also wish to (iii) explore pharmacists views on the interventions

Data from this pilot will enable the investigators to determine whether a larger multisite study is feasible. The aims of a larger study being to determine if either of the two interventions being tested result in an increased proportion of women using effective ongoing contraception compared to the control.

DETAILED DESCRIPTION:
The investigators propose to test 2 pharmacy based interventions to increase uptake of effective contraception after EC:

1. Pharmacists would provide one packet of progestogen-only pills to women, so that they would have 28 days to arrange an appointment with contraceptive services to get a supply of ongoing contraception.
2. Rapid access to a family planning clinic upon presentation of their empty(used) packet of EC. Women would be seen as a 'walk-in' (without appointment) and ongoing contraception discussed and provided.

These interventions would be compared with the status quo, i.e. pharmacists give verbal advice and written information on local contraceptive services where ongoing contraception can be accessed.

The interventions that we are testing are low cost i.e one packet of progestogen-only pills (£3 for most costly brand) plus additional consultation time with the pharmacist (estimated 20 mins@ £1 per minute), versus the staff consultation time in a family planning clinic. In the family planning clinic, women would be seen as a 'walk-in' and so this may not add costs, since staff are already present.These interventions could, if shown to be effective, offer huge costs savings to the NHS, by reducing the costs of unintended pregnancies (abortion, miscarriage, birth).

ELIGIBILITY:
Inclusion Criteria:

* age >= 16 yrs
* requesting emergency contraception
* eligible for emergency contraception
* written , informed consent

Exclusion Criteria:

* age < 16 yrs
* not able to give written , informed consent

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 168 (Actual)
Dates: Start 2012-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon T Cameron, MBChB, Principal Investigator — University of Edinburgh
Locations (1):
- Chalmers sexual and reproductive health service, Edinburgh, Lothian, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from end April 2012 - end December 2012 (8 month period). Recruitment of participants by community pharmacists within 11 community pharmacies in Edinburgh.
  All participating pharmacists trained by the research team prior to commencing recruitment of participants.
Groups:
- Rapid Access: rapid access to family planning service
  rapid access to contraceptive service
Period: Overall Study
Arm/Group | Control (Standard Care) | Rapid Access | Progestogen Only Pill
Started | 54 (54 participants recruited to this arm) | 58 (58 participants recruited to this arm) | 56 (56 participants recruited to this arm)
Completed | 35 (35 participants successfully contacted to complete telephone follow-up at 6-8 weeks.) | 28 (28 participants successfully contacted to complete telephone follow-up at 6-8 weeks.) | 39 (39 participants successfully contacted to complete telephone follow-up at 6-8 weeks.)
Not Completed | 19 | 30 | 17
Not completed — Lost to Follow-up | 19 | 30 | 17

BASELINE CHARACTERISTICS:
Population: Baseline analysis conducted on all participants successfully contacted for telephone follow-up at 6-8weeks post enrollment to study. no baseline analysis possible on those recruited in pharmacy but lost to follow-up.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control (Standard Care) | Rapid Access | Progestogen Only Pill | Total
Number analyzed (Participants) | 35 | 28 | 39 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 23 (4.5) | 25 (5.6) | 22 (5.2) | 23 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 28 | 39 | 102
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 35 | 28 | 39 | 102
Contraception use at time of enrollment [Number; unit: participants]
  None | 12 | 8 | 13 | 33
  Condoms | 19 | 17 | 26 | 62
  Other method | 4 | 3 | 0 | 7

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Uptake of Effective Ongoing Contraception (Not Condoms)
Description: Outcome measure identified when participants conducted for agreed telephone interview 6-8 weeks following recruitment to study. Participants asked via telephone what method of contraception, if any, there were currently using.
Time Frame: 6-8 weeks after EC
Population: A small number of participants were identified who had been recruited to the study although were already using an effective method of contraception (i.e. using a contraceptive pill but had forgot to take), and continued to use the same method at follow-up. These participants were excluded from analysis.
Measure: Number; unit: participants
Arm/Group | Control (Standard Care) | Rapid Access | Progestogen Only Pill
Number analyzed (Participants) | 31 | 25 | 39
participants
  Effective contraception | 5 | 13 | 22
  Long acting contraception | 0 | 5 | 3
  No contraception / barrier method | 26 | 12 | 17
Statistical Analysis 1: Comparison: Control (Standard Care) vs Progestogen Only Pill; Cluster randomised study design - statisitical analysis takes this into account. Analaysis was conducted at a cluster level and the proportions in each cluster using effective contraception were compared between groups by 2-sample t tests, weighted by the different number of patients in each cluster. Comparison of number of women using effective contraception at 6-8 weeks in progestogen only pill group compared to control; Test type: Superiority or Other; p < 0.001, t-test, 2 sided; see above description of analysis taking into account cluster randomisation; relative probability = 3.13, 95% CI [1.90 to 5.13]
Statistical Analysis 2: Comparison: Control (Standard Care) vs Rapid Access; Cluster randomised study design - statisitical analysis takes this into account. Analaysis was conducted at a cluster level and the proportions in each cluster using effective contraception were compared between groups by 2-sample t tests, weighted by the different number of patients in each cluster. Comparison of number of women using effective contraception at 6-8 weeks in rapid access group compared to control; Test type: Superiority or Other; p = 0.006, t-test, 2 sided — see above comments regarding analysis taking cluster randomised account into consideration; relative probability = 2.57, 95% CI [1.55 to 4.27]

2. Secondary Outcome: Pharmacy Recruitment Rates
Description: Proportion of participants that pharmacists were successful in recruiting during the specified 8 month recruitment time period. Initial target set to recruit 60 participants to each arm/group.
Time Frame: 8 months
Measure: Number; unit: participants
Arm/Group | Control (Standard Care) | Rapid Access | Progestogen Only Pill
Number analyzed (Participants) | 60 | 60 | 60
participants
  Recruited | 54 | 58 | 56
  Not recruited from target figure | 6 | 2 | 4

3. Secondary Outcome: Completeness (Quality) of Data Recorded by Pharmacists (Numbers of Women Attending for EC,Demographics of All Attendees- Age, Ethnicity Etc)
Time Frame: 8 months
Reporting Status: Not Posted

4. Secondary Outcome: Proportion of Women Who Agree to Participate Who Can be Successfully Contacted
Time Frame: 8 months
Measure: Number; unit: participants
Arm/Group | Control (Standard Care) | Rapid Access | Progestogen Only Pill
Number analyzed (Participants) | 54 | 58 | 56
participants
  Women successfully contacted for follow-up | 35 | 28 | 39
  Not contacted / lost to follow-up | 19 | 30 | 17

5. Other Pre Specified Outcome: Qualitative Outcomes : Women's Views on Different Measures to Determine Validity of Self-reported Data on Contraceptive Use , Determined by in Depth Interviews.
Time Frame: 8 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Qualitative Outcomes : Pharmacist's Views on Interventions and Any Study Difficulties
Time Frame: 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 14 months
Arm/Group | Control (Standard Care) | Rapid Access | Progestogen Only Pill
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/58 | 0/56
Other Adverse Events (participants affected / at risk) | 0/54 | 0/58 | 0/56

LIMITATIONS AND CAVEATS:
Loss to follow-up relatively high. Self-reporting of primary outcome measure (contraceptive method at time of follow-up). Would have been preferable to be able to validate this.

Pharmacists unable to record demographic data of those not recruited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No